CLINICAL TRIAL: NCT02329366
Title: Development of a Cellular Biomarker for the Diagnosis and Treatment of Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 14328
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Foot Ulcer; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2 | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In this study, diabetic patients undergoing Diabetic Foot Ulcer debridement under the standard of care will be asked for their permission to collect the debrided tissue for use in scientific research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic Foot Ulcer Group: Subjects in this group will have tissue specimens collected from their Diabetic Foot Ulcer during Standard of Care debridement.
  Interventions: Other: Specimen Collection
- Control Group: Skin tissue samples will be collected from subjects undergoing routine surgical procedures during which normal skin is removed
  Interventions: Other: Specimen Collection

INTERVENTIONS:
Other: Specimen Collection — . In this study, diabetic patients undergoing DFU debridement under the standard of care will be asked for their permission to collect the debrided tissue for use in scientific research.

SUMMARY:
This project aims to result in the identification of such markers, and the development of a feasible quantitative method of distinguishing between tissue that has the capacity to heal and tissue that does not, thus identifying a non-healing phenotype.

DETAILED DESCRIPTION:
The goal of this project is to identify objective, quantitative biological and molecular markers that correlate with healing outcomes for diabetic foot ulcers (DFUs) using debrided tissue of patients with wounds. This project aims to result in the identification of such markers, and the development of a feasible quantitative method of distinguishing between tissue that has the capacity to heal and tissue that does not, thus identifying a non-healing phenotype. The ability to differentiate between healing and non-healing tissue at the onset of wound care will allow for the use of targeted therapies and earlier initiation of aggressive treatments where indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18
* Type 2 Diabetes
* A break in the skin on the foot ≥ 0.5cm2 and is Grade 1 or 2 as defined by the Wagner grading system
* Hemoglobin A1c ≥ 5.9%
* Ability to provide written informed consent

Exclusion Criteria:

* Any experimental drugs taken orally or topically within 4 weeks of study entry
* Malignant disease at/or in proximity to the DFU
* Target wound of malignant origin
* Failure to satisfy at least one inclusion criterion for one of the two study groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both male and female patients at Winthrop University Hospital over the age of 18 with Type 2 Diabetes and a Diabetic Foot Ulcer are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
To identify objective, quantitative biological and molecular markers that correlate with healing outcomes for diabetic foot ulcers (DFUs) using debrided tissue of patients with wounds | Undetermined

CONTACTS AND LOCATIONS:
Overall Officials: Harold Brem, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States